CLINICAL TRIAL: NCT01371734
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study To Evaluate The Efficacy, Safety And Tolerability Of Desvenlafaxine Succinate Sustained-release (Dvs Sr) In The Treatment Of Children And Adolescent Outpatients With Major Depressive Disorder
Brief Title: A Study Of DVS SR In Treatment Of Children And Adolescent Outpatients With MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2061032; 3151A6-3343 (Other: Alias Study Number); 2008-001875-32 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Arm 1 - high dose (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release
- Experimental Arm 2 - low dose (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release — Subjects randomized to DVS SR treatment arm will receive 25, 35, or 50 mg/day based on subject weight at the Baseline visit.
  Arms: Experimental Arm 1 - high dose
Drug: Desvenlafaxine Succinate Sustained-Release — Subjects randomized to DVS SR treatment arm will receive 20, 25, or 35 mg/day based on subject weight at the Baseline visit.
  Arms: Experimental Arm 2 - low dose
Drug: Placebo — Subjects randomized to the Placebo treatment arm will receive placebo tablets
  Arms: Placebo Arm

SUMMARY:
This is a double-blind study evaluating Desvenlafaxine Succinate Sustained-Release (DVS SR) versus placebo in the Treatment of Children and Adolescent Outpatients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Age >=7 and <18 years of age
* Primary diagnosis of major depressive disorder (MDD)
* CDRS-R score >40

Exclusion Criteria:

* History of suicidal behavior or requires precaution against suicide
* Not in generally healthy medical condition
* History of psychosis or bipolar disorder
* Seizure disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 363 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (39):
  - Children's Hospital of Alabama Laboratory, Birmingham, Alabama
  - The University of Alabama at Birmingham, Office of Psychiatric Research, Birmingham, Alabama
  - Center for Advanced Improvement, Tucson, Arizona
  - Sun Valley Research Center, Imperial, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Bliss Basement Pharmacy - Hartford Hospital, Hartford, Connecticut
  - Institute of Living/Hartford Hospital, Hartford, Connecticut
  - Institute of Living, Hartford, Connecticut
  - SJS Clinical Research, Inc., Destin, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Millenia Psychiatry & Research, Inc., Orlando, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - Clinco, Terre Haute, Indiana
  - Louisiana State University Health Sciences Center-Psychopharmacology Research Clinic, Shreveport, Louisiana
  - Drug:University Health Shreveport Outpatient, Shreveport, Louisiana
  - Pharmasite Research Inc, Baltimore, Maryland
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Erie County Medical Center / State University of New York at Buffalo affiliate, Buffalo, New York
  - The Zucker Hillside Hospital, North Shore-Long Island Jewish Health System, Glen Oaks, New York
  - Bioscience Research, LLC., Mount Kisco, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Stony Brook University Medical Center, Child And Adolescent Psychiatry, Stony Brook, New York
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Discovery and Wellness Center for Children/University Hospitals Case Medical Center, Cleveland, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Research Strategies of Memphis, LLC., Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Alliance Research Group, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Treatment Center, Richmond, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
- Chile (2):
  - Biomedica Research Group, Santiago, Santiago Metropolitan
  - Optima Salud, Santiago, Santiago Metropolitan
- Hospital Universitario Dr. Jose Eleuterio Gonzalez, Departamento de Psiquiatria, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Derived] Atkinson S, Lubaczewski S, Ramaker S, England RD, Wajsbrot DB, Abbas R, Findling RL. Desvenlafaxine Versus Placebo in the Treatment of Children and Adolescents with Major Depressive Disorder. J Child Adolesc Psychopharmacol. 2018 Feb;28(1):55-65. doi: 10.1089/cap.2017.0099. Epub 2017 Nov 29. PMID 29185786
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061032&StudyName=A%20Study%20Of%20DVS%20SR%20In%20Treatment%20Of%20Children%20And%20Adolescent%20Outpatients%20With%20MDD

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matched placebo tablets administered once daily for 8 weeks (treatment phase), followed by placebo tablets administered once daily for 1 week (taper phase) only for those participants not entering the extension study.
- DVS SR Low Dose: DVS SR tablets 10 or 20 mg (based on weight at the baseline visit) administered once daily for the first week of treatment (titration phase) then 20, 25 or 35 mg (based on weight at the baseline visit) administered once daily for the next 7 weeks of treatment, followed by 10 or 20 mg (based on weight at the baseline visit) administered once daily for 1 week (taper phase) only for those participants not entering the extension study.
- DVS SR High Dose: DVS SR tablets 10 or 20 mg (based on weight at the baseline visit) administered once daily for the first week of treatment (titration phase) then 25, 35 or 50 mg (based on weight at the baseline visit) administered once daily for the next 7 weeks of treatment, followed by 10 or 20 mg (based on weight at the baseline visit) administered once daily for 1 week (taper phase) only for those participants not entering the extension study.
Period: Overall Study
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Started | 120 | 122 | 121
Completed | 97 | 103 | 104
Not Completed | 23 | 19 | 17
Not completed — Other | 2 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 9
Not completed — Lost to Follow-up | 5 | 3 | 1
Not completed — Protocol Violation | 3 | 1 | 2
Not completed — Adverse Event | 8 | 8 | 3
Not completed — Lack of Efficacy | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population - included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose | Total
Number analyzed (Participants) | 120 | 122 | 121 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.2 (2.68) | 13.1 (2.80) | 12.9 (3.01) | 13.0 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 69 | 76 | 205
  Male | 60 | 53 | 45 | 158

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Children's Depression Rating Scale, Revised (CDRS-R) Total Score (n=102, 104, 106)
Description: Clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment). Total score calculated as sum of the 17 items (range 1 to 119); higher score indicates greater impairment. Mean change from baseline was adjusted for the baseline total score, age group and gender.
Time Frame: Baseline and Week 8
Population: Intention-To-Treat (ITT) Population - included all randomized participants who received at least 1 dose of study drug, had a baseline primary efficacy assessment, and had at least one post-baseline primary efficacy assessment.
  n is the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Number analyzed (Participants) | 119 | 120 | 121
Score on a scale | -22.85 (1.13) | -23.70 (1.12) | -24.37 (1.12)
Statistical Analysis 1: Comparison: Placebo vs DVS SR Low Dose; Adjusted mean difference = Placebo - DVS SR Low Dose; Test type: Superiority or Other; p = 0.587, Mixed-effects model for repeated measure; Hochberg procedure was used to control for multiplicity; Mean Difference (Net) = 0.85, 95% CI 2-sided [-2.23 to 3.94]
Statistical Analysis 2: Comparison: Placebo vs DVS SR High Dose; Adjusted mean difference = Placebo - DVS SR High Dose; Test type: Superiority or Other; p = 0.333, Mixed-effects model for repeated measure; Hochberg procedure was used to control for multiplicity; Mean Difference (Net) = 1.52, 95% CI 2-sided [-1.56 to 4.61]

2. Secondary Outcome: Change From Baseline to Week 8 in the Clinical Global Impression of Severity (CGI-S) Score (n=102, 105, 106)
Description: A 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline. Mean change from baseline was adjusted for the baseline total score, age group and gender.
Time Frame: Baseline and Week 8
Population: ITT Population n is the number of participants with evaluable data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Number analyzed (Participants) | 119 | 120 | 121
Score on a scale | -1.49 (0.11) | -1.51 (0.11) | -1.65 (0.11)
Statistical Analysis 1: Comparison: Placebo vs DVS SR Low Dose; Adjusted mean difference = Placebo - DVS SR Low Dose; Test type: Superiority or Other; p = 0.923, Mixed-effects model for repeated measure; Hochberg procedure was used to control for multiplicity; Mean Difference (Net) = 0.015, 95% CI 2-sided [-0.29 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs DVS SR High Dose; Adjusted mean difference = Placebo - DVS SR High Dose; Test type: Superiority or Other; p = 0.302, Mixed-effects model for repeated measure; Hochberg procedure was used to control for multiplicity; Mean Difference (Net) = 0.161, 95% CI 2-sided [-0.14 to 0.47]

3. Secondary Outcome: Percentage of Participants by Clinical Global Impression Improvement (CGI-I) Score at Weeks 1, 2, 3, 4, 6, and 8
Description: A 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score equals (=) more affected.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: ITT Population n is the number of participants with non-missing values
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Number analyzed (Participants) | 119 | 120 | 121
Percentage of Participants
  Week 1, Very Much Improved (n=113, 112,115) | 2.7 | 0.9 | 2.6
  Week 1, Much Improved (n=113, 112, 115) | 6.2 | 9.8 | 12.2
  Week 1, Minimally Improved (n=113, 112, 115) | 38.9 | 37.5 | 33.9
  Week 1, No Change (n=113, 112, 115) | 49.6 | 51.8 | 46.1
  Week 1, Minimally Worse (n=113, 112, 115) | 2.7 | 0 | 5.2
  Week 1, Much Worse (n=113, 112, 115) | 0 | 0 | 0
  Week 1, Very Much Worse (n=113, 112, 115) | 0 | 0 | 0
  Week 2, Very Much Improved (n=114, 115, 109) | 4.4 | 6.1 | 10.1
  Week 2, Much Improved (n=114, 115, 109) | 26.3 | 26.1 | 23.9
  Week 2, Minimally Improved (n=114, 115, 109) | 36.8 | 38.3 | 35.8
  Week 2, No Change (n=114, 115, 109) | 31.6 | 25.2 | 29.4
  Week 2, Minimally Worse (n=114, 115, 109) | 0 | 4.3 | 0
  Week 2, Much Worse (n=114, 115, 109) | 0.9 | 0 | 0.9
  Week 2, Very Much Worse (n=114, 115, 109) | 0 | 0 | 0
  Week 3, Very Much Improved (n=108, 110, 110) | 10.2 | 10.9 | 18.2
  Week 3, Much Improved (n=108, 110, 110) | 20.4 | 26.4 | 24.5
  Week 3, Minimally Improved (n=108, 110, 110) | 47.2 | 44.5 | 35.5
  Week 3, No Change (n=108, 110, 110) | 20.4 | 15.5 | 21.8
  Week 3, Minimally Worse (n=108, 110, 110) | 1.9 | 1.8 | 0
  Week 3, Much Worse (n=108, 110, 110) | 0 | 0 | 0
  Week 3, Very Much Worse (n=108, 110, 110) | 0 | 0.9 | 0
  Week 4, Very Much Improved (n=104,108,113) | 14.4 | 17.6 | 15.0
  Week 4, Much Improved (n=104,108,113) | 30.8 | 36.1 | 31.0
  Week 4, Minimally Improved (n=104,108,113) | 35.6 | 30.6 | 35.4
  Week 4, No Change (n=104,108,113) | 19.2 | 14.8 | 17.7
  Week 4, Minimally Worse (n=104,108,113) | 0 | 0.9 | 0.9
  Week 4, Much Worse (n=104,108,113) | 0 | 0 | 0
  Week 4, Very Much Worse (n=104,108,113) | 0 | 0 | 0
  Week 6, Very Much Improved (n=106,104,104) | 19.8 | 20.2 | 26.9
  Week 6, Much Improved (n=106,104,104) | 29.2 | 36.5 | 24.0
  Week 6, Minimally Improved (n=106,104,104) | 31.1 | 24.0 | 31.7
  Week 6, No Change (n=106,104,104) | 16.0 | 14.4 | 14.4
  Week 6, Minimally Worse (n=106,104,104) | 2.8 | 2.9 | 1.9
  Week 6, Much Worse (n=106,104,104) | 0 | 1.9 | 1.0
  Week 6, Very Much Worse (n=106,104,104) | 0.9 | 0 | 0
  Week 8, Very Much Improved (n=102,105,106) | 21.6 | 19.0 | 25.5
  Week 8, Much Improved (n=102,105,106) | 34.3 | 37.1 | 36.8
  Week 8, Minimally Improved (n=102,105,106) | 28.4 | 24.8 | 21.7
  Week 8, No Change (n=102,105,106) | 15.7 | 18.1 | 15.1
  Week 8, Minimally Worse (n=102,105,106) | 0 | 1.0 | 0.9
  Week 8, Much Worse (n=102,105,106) | 0 | 0 | 0
  Week 8, Very Much Worse (n=102,105,106) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs DVS SR Low Dose; Week 1; Test type: Superiority or Other; p = 0.729, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs DVS SR High Dose; Week 1; Test type: Superiority or Other; p = 0.756, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs DVS SR Low Dose; Week 2; Test type: Superiority or Other; p = 0.765, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs DVS SR High Dose; Week 2; Test type: Superiority or Other; p = 0.475, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs DVS SR Low Dose; Week 3; Test type: Superiority or Other; p = 0.310, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs DVS SR High Dose; Week 3; Test type: Superiority or Other; p = 0.105, Chi-squared, Corrected
Statistical Analysis 7: Comparison: Placebo vs DVS SR Low Dose; Week 4; Test type: Superiority or Other; p = 0.254, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs DVS SR High Dose; Week 4; Test type: Superiority or Other; p = 0.887, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs DVS SR Low Dose; Week 6; Test type: Superiority or Other; p = 0.475, Cochran-Mantel-Haenszel
Statistical Analysis 10: Comparison: Placebo vs DVS SR High Dose; Week 6; Test type: Superiority or Other; p = 0.407, Cochran-Mantel-Haenszel
Statistical Analysis 11: Comparison: Placebo vs DVS SR Low Dose; Week 8; Test type: Superiority or Other; p = 0.696, Cochran-Mantel-Haenszel
Statistical Analysis 12: Comparison: Placebo vs DVS SR High Dose; Week 8; Test type: Superiority or Other; p = 0.462, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With a CGI-I Response Defined as a Score of 'Very Much Improved' or 'Much Improved'
Description: A 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale. Higher score = more affected.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: ITT Population n is the number of participants with non-missing values
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Number analyzed (Participants) | 119 | 120 | 121
Percentage of Participants
  Week 1 (n=113, 112, 115) | 8.85 | 10.71 | 14.78
  Week 2 (n=114, 115, 109) | 30.70 | 32.17 | 33.94
  Week 3 (n=108, 110, 110) | 30.56 | 37.27 | 42.73
  Week 4 (n=104, 108, 113) | 45.19 | 53.70 | 46.02
  Week 6 (n=106, 104, 104) | 49.06 | 56.73 | 50.96
  Week 8 (n=102, 105, 106) | 55.88 | 56.19 | 62.26
Statistical Analysis 1: Comparison: Placebo vs DVS SR Low Dose; Week 1; Test type: Superiority or Other; p = 0.633, Regression, Logistic; Odds Ratio (OR) = 0.806, 95% CI 2-sided [0.333 to 1.951]
Statistical Analysis 2: Comparison: Placebo vs DVS SR High Dose; Week 1; Test type: Superiority or Other; p = 0.172, Regression, Logistic; Odds Ratio (OR) = 0.561, 95% CI 2-sided [0.245 to 1.285]
Statistical Analysis 3: Comparison: Placebo vs DVS SR Low Dose; Week 2; Test type: Superiority or Other; p = 0.826, Regression, Logistic; Odds Ratio (OR) = 0.939, 95% CI 2-sided [0.536 to 1.644]
Statistical Analysis 4: Comparison: Placebo vs DVS SR High Dose; Week 2; Test type: Superiority or Other; p = 0.599, Regression, Logistic; Odds Ratio (OR) = 0.860, 95% CI 2-sided [0.489 to 1.511]
Statistical Analysis 5: Comparison: Placebo vs DVS SR Low Dose; Week 3; Test type: Superiority or Other; p = 0.248, Regression, Logistic; Odds Ratio (OR) = 0.713, 95% CI 2-sided [0.402 to 1.265]
Statistical Analysis 6: Comparison: Placebo vs DVS SR High Dose; Week 3; Test type: Superiority or Other; p = 0.048, Regression, Logistic; Odds Ratio (OR) = 0.564, 95% CI 2-sided [0.320 to 0.995]
Statistical Analysis 7: Comparison: Placebo vs DVS SR Low Dose; Week 4; Test type: Superiority or Other; p = 0.210, Regression, Logistic; Odds Ratio (OR) = 0.708, 95% CI 2-sided [0.412 to 1.216]
Statistical Analysis 8: Comparison: Placebo vs DVS SR High Dose; Week 4; Test type: Superiority or Other; p = 0.893, Regression, Logistic; Odds Ratio (OR) = 0.964, 95% CI 2-sided [0.564 to 1.646]
Statistical Analysis 9: Comparison: Placebo vs DVS SR Low Dose; Week 6; Test type: Superiority or Other; p = 0.228, Regression, Logistic; Odds Ratio (OR) = 0.714, 95% CI 2-sided [0.413 to 1.235]
Statistical Analysis 10: Comparison: Placebo vs DVS SR High Dose; Week 6; Test type: Superiority or Other; p = 0.751, Regression, Logistic; Odds Ratio (OR) = 0.916, 95% CI 2-sided [0.531 to 1.579]
Statistical Analysis 11: Comparison: Placebo vs DVS SR Low Dose; Week 8; Test type: Superiority or Other; p = 0.925, Regression, Logistic; Odds Ratio (OR) = 0.974, 95% CI 2-sided [0.561 to 1.689]
Statistical Analysis 12: Comparison: Placebo vs DVS SR High Dose; Week 8; Test type: Superiority or Other; p = 0.342, Regression, Logistic; Odds Ratio (OR) = 0.764, 95% CI 2-sided [0.438 to 1.331]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from informed consent and assent through the first follow up visit (Week 11) for non-serious AEs; the second follow up visit (Week 13) for serious AEs (SAEs); or at Week 8 for participants entering the extension study.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | DVS SR Low Dose | DVS SR High Dose
Serious Adverse Events (participants affected / at risk) | 2/120 | 2/122 | 1/121
Other Adverse Events (participants affected / at risk) | 34/120 | 46/122 | 53/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | DVS SR Low Dose (N=122) | DVS SR High Dose (N=121)
Abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | DVS SR Low Dose (N=122) | DVS SR High Dose (N=121)
Abdominal pain upper (Gastrointestinal disorders) | 9 | 7 | 11
Nausea (Gastrointestinal disorders) | 7 | 12 | 14
Vomiting (Gastrointestinal disorders) | 4 | 1 | 9
Fatigue (General disorders) | 2 | 4 | 9
Nasopharyngitis (Infections and infestations) | 2 | 8 | 7
Headache (Nervous system disorders) | 15 | 22 | 25
Insomnia (Psychiatric disorders) | 1 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less